CLINICAL TRIAL: NCT00725556
Title: The Development of Autistic Children Based on Mother´s Response in Autism Behavior Checklist
Brief Title: The Development of Autistic Children Based on Mothers´Response in Autism Behavior Checklist
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Ana Carina Tamanaha, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ana Carina Tamanaha
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Autism; Asperger Syndrome
Keywords: Autism; Asperger Syndrome
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Speech therapy
  Interventions: Other: Speech Therapy

INTERVENTIONS:
Other: Speech Therapy — Speech Therapy

SUMMARY:
The purpose of this study is to evaluate the process of development of autistic children, in a direct and indirect intervention context from mother´s response in Autism Behavior Checklist.

DETAILED DESCRIPTION:
Aim: We evaluated the process of development of autistic children, in a direct and indirect intervention context from mother´s response in Autism Behavior Checklist.

Method:

The sample were composed of 11 mothers of children diagnosed with Autism (6) and Asperger Syndrome (5), according to the criteria established by the DSM IVtr (APA, 2002). These children were randomly divided into two groups: Six were receiving both direct and indirect intervention (Therapy Group -TG), and five were receiving exclusively indirect intervention (Orientation Group - OG). We used the Autism Behavior Checklist (Krug et al., 1993), adapted to Portuguese on three occasions: at the beginning, six months later and 12 months later. This is a list of nonadaptive behaviors (57), in the areas: Sensorial, Body and Object Use, Language, Social and Relating.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Autism or Asperger Syndrome
* Age (children)
* Adherence in the study (at least 70%)

Exclusion Criteria:

* Others clinical diagnosis

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the process of development of autistic children, in a direct and indirect intervention context from mother´s response in Autism Behavior Checklist. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carina Tamanaha, Student, Principal Investigator — Federal University of São Paulo
Locations (1):
- Ana Carina Tamanaha, São Paulo, São Paulo, Brazil